CLINICAL TRIAL: NCT02919202
Title: A Randomised Controlled Trial Investigating a Comparison of Fluoride Varnish vs Self-Etching Dentine Bonding Agent in the Reduction of Cervical Dentine Sensitivity in Patients Attending a General Dental Practice in West Sussex, UK.
Brief Title: Clinical Trial to Compare the Efficacy of a Fluoride Gel and a Dental Bonding Agent in Treatment of Tooth Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ResGov 354
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoride Varnish (Experimental): Colgate Fluoride Varnish Suspension. 2.26% Sodium Fluoride.
  Interventions: Procedure: Colgate Fluoride Varnish Suspension. 2.26% Sodium Fluoride.
- SEDBA (Active Comparator): Self-etching Dentine Bonding Agent. Scotchbond Universal by 3M ESPE. Topical application followed by light curing for 20 seconds.
  Interventions: Procedure: Self-etching Dentine Bonding Agent

INTERVENTIONS:
Procedure: Colgate Fluoride Varnish Suspension. 2.26% Sodium Fluoride. — Topical application to exposed dentine on one occasion.
  Other Names: Duraphat Varnish
  Arms: Fluoride Varnish
Procedure: Self-etching Dentine Bonding Agent — Topical application to exposed dentine on one occasion followed by light-curing procedure.
  Other Names: Scotchbond Universal
  Arms: SEDBA

SUMMARY:
This study compares the efficacy of two dental interventions in the treatment of cervical dentine sensitivity. The participants will be selected from adult dental patients registered at a general dental practice in West Sussex, UK. The participants will be split into 2 groups. One group will receive the intervention of topical fluoride varnish application while the other group will receive a topical application of self-etching dentine bonding agent.

DETAILED DESCRIPTION:
Topical Fluoride Varnish(TFV) and Self-Etching Dentine Bonding Agent (SEDBA) are both routinely used in dentistry in the management of cervical dentine sensitivity(CDS). Both interventions are topically applied and well tolerated by patients. The interventions differ in mechanism of action. TFV releases fluoride which is incorporated into the organic matrix of dentine making the dentine tubules less conductive. Dentinal tubules form the key conduit between stimulus and pain perception in the tooth. SEDBA differs in that it penetrates and occludes the tubules. It is light cured for an almost instant set time.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60.
* Exhibiting CDS elicited by the two test stimuli in relation at least one tooth.

Exclusion Criteria:

* Patients who have undergone comprehensive periodontal treatment in the past 3 months.
* Patients under the age of 18 or unable to provide valid consent.
* Teeth that have visible fracture lines, caries, crowns or have been endodontically treated.
* Patients taking analgesic medication for any systemic conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 14 days
  to measure pain/sensitivity perception

CONTACTS AND LOCATIONS:
Overall Officials: Claire Parkin, PhD, Principal Investigator — University of Kent
Locations (1):
- Carfax Dental Practice, Horsham, West Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No